CLINICAL TRIAL: NCT05297617
Title: Single-arm Study to De-escalate Adjuvant Endocrine Therapy Duration in Women With HR+ HER2- Breast Cancer at Very Low Risk of Metastasis
Brief Title: Deescalation of Endocrine Therapy Duration in Women With HR+ HER2- Breast Cancer at Very Low Risk
Acronym: LESS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Agendia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2103; 2021-002889-41 (EudraCT Number); 2024-514480-26-00 (EU CTIS Number)
Record Dates: First submitted 2022-03-16; First posted 2022-03-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, national, multicenter, single-arm, interventional, non-threshold crossing phase II study evaluating a therapeutic de-escalation that limits adjuvant hormone therapy to 2 years of aromatase inhibitor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aromatase inhibitor (Experimental): Patient will receive standard endocrine therapy (single agent aromatase inhibitors) for a maximum of 2 years.
  Interventions: Drug: Anti-aromatase inhibitor

INTERVENTIONS:
Drug: Anti-aromatase inhibitor — Treatment will be either:
  * Letrozole, given per os, 2.5 mg daily
  * Anastrozole, given per os, 1 mg daily
  * Exemestane, given per os, 25 mg daily

SUMMARY:
Hormone therapy is recommended for five years in all patients with hormone receptor-positive breast cancer, but there is no consensus on its duration in low-risk tumours and especially in postmenopausal women. Adjuvant endocrine therapy (ET) is associated with substantial side effects and long-term decreased quality of life.

Moreover, while it has been shown that ET provides a real benefit in reducing the relapse rate over time, the deterioration in quality of life may also have a negative effect on patient adherence to treatment. It is therefore important to offer treatment to women with low-risk cancer less intensive treatment strategies. If recent trials tested longer durations as compared to 5 years for high-risk cancers, older trials have tested shorter durations. The 5-year duration appeared at that time as the gold standard because of optimal benefit-risk ratios of tamoxifen among high-risk patients. However shorter treatments of 2-3 years were already associated with substantial benefits and may be enough for very low risk patients.

DETAILED DESCRIPTION:
Adjuvant ET is the cornerstone treatment of localized hormone-receptor positive breast cancer, with demonstrated benefits on overall survival (30-40% relative decrease in mortality) but also on the risk of local and contralateral relapse (43-50% relative decrease). While the relative benefit of 5 years ET is identical for small tumors as compared to larger ones, the absolute benefit is much lower, and the risk-benefit ratio may therefore become very questionable given the frequent and impactful side effects of ET. If recent trials tested longer durations as compared to 5 years for high-risk cancers, older trials have tested shorter durations. Five years appeared at that time as the gold standard because of optimal benefit-risk ratios of tamoxifen among rather high-risk patients. However shorter treatments of 2-3 years were already associated with substantial benefits and may be enough for very low risk patients. The purpose of this study is to demonstrate that adjuvant hormone therapy limited to 2 years of antiaromatase in postmenopausal women with a good prognosis can ensure very high survival without metastatic relapse and allows a reduction of side effects and a better quality of life. The 5-year DMFS was excellent in patients with low risk Luminal A tumors who received endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women: Postmenopausal status is defined by any of the following:

   * Prior bilateral oophorectomy
   * Age ≥60 years
   * Age >50 and <60 years and amenorrheic for at least 12 months, and follicle-stimulating hormone (FSH) and estradiol in the postmenopausal range
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
3. Women with histologically proven invasive unilateral breast cancer Note: In case of a multifocal invasive tumor, all lesions (maximum 3 infiltrating lesions allowed) must be of identical phenotype and low biological risk
4. M0: Not clinically nor radiologically detectable metastases at time of inclusion
5. Primary tumor completely resected and adequate axillary surgery performed, according to current standards
6. IHC expression of the estrogen receptor and/or progesterone receptor ≥50%
7. HER2 negative according to ASCO criteria in immunohistochemistry and/or genomic analysis (HER2 negativity is defined as IHC 0-1+, or [IHC 2+ and FISH or CISH nonamplified])
8. No indication of adjuvant chemotherapy
9. pT1 (tumor ≤20 mm), pN0, Grade 1 or Grade 2 OR pT2 (tumor ≤30 mm) and pN0, Grade 1 or Grade 2

   Note 1: patient with Grade 2 pT2pN0 tumor must be aged under 70 years of age and should receive a genomic test as part of standard care (RIHN reimbursement)
10. Patient considered has having a luminal A ultralow risk of metastatic recurrence (i.e.less than 5% risk of metastatic relapse at 10 years) according to MammaPrint® and Blueprint® tests.

    Note 1: To be eligible, MammaPrint index score should be > +0.355
11. Patients eligible to receive or have recently started (with a maximum of 4 months of adjuvant hormone therapy prior to enrollment) an adjuvant hormone therapy (letrozole, anastrozole, or exemestane)
12. Patient is willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures
13. Patients must be affiliated to a Social Security System (or equivalent)
14. Patient must have signed a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.

Exclusion Criteria:

1. Patients who received a neo-adjuvant hormone therapy, a neo-adjuvant or adjuvant chemotherapy or preoperative medical treatment
2. Any local or regional recurrence or metastatic disease
3. Non-invasive carcinoma
4. Bilateral breast cancer (except in case of contralateral DCIS), or history of other invasive ipsi- or contralateral breast cancer
5. Patients with a history of another malignancy, except for properly treated cervical carcinoma in situ, and non-melanoma cancer of the skin
6. Women with high-risk breast cancer predisposing deleterious germline mutations
7. Contra-indications to the administration of anti-aromatase inhibitors
8. Patients enrolled in another therapeutic study within 30 days prior to inclusion
9. Patients with any other disease or illness, which requires hospitalization or is incompatible with the trial treatment
10. Patients unwilling or unable to comply with trial obligations for geographic, social, physical or psychological reasons, or who are unable to understand the purpose and procedures of the trial
11. Persons deprived of their liberty or under protective custody or guardianship

Min Age: 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2030-11-12 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Distant relapse-free interval (DRFI) | From date of beginning of hormonotherapy to onset of metastases or death, up to 5-years.
  Distant relapse-free interval (DRFI) is defined as the time from date of beginning of hormonotherapy to the date of first event of distant recurrence or breast cancer related death

SECONDARY OUTCOMES:
Distant Disease-Free Survival (DDFS) | From date of beginning of hormonotherapy to the date of first event of distant recurrence, death from any cause or secondary non-breast cancer up to 10 years
  DDFS is defined as the time from date of beginning of hormonotherapy to the date of first event of distant recurrence, death from any cause or secondary non-breast cancer.
Invasive disease free survival (iDFS) | From date of beginning of hormonotherapy to onset of invasive event, second cancer, or death, up to 10 years.
  Invasive disease free survival is defined as duration of time from date of registration until first appearance of invasive local, regional, or distant recurrence (including invasive ipsilateral breast cancer recurrence), invasive contralateral breast cancer, second primary non breast invasive cancer (excluding non-melanoma skin cancer), or death from any cause.
Invasive breast cancer-free survival (iBCFS) | From date of beginning of hormonotherapy to onset of invasive event or death, up to 10 years.
  Invasive disease free survival is defined as the delay between date of inclusion and first appearance of invasive local, regional, or distant recurrence (including invasive ipsilateral breast cancer recurrence), invasive contralateral breast cancer, or death from any cause.
Breast cancer-specific survival (BCSS) | From date of beginning of hormonotherapy to death from breast cancer, up to 10 years.
  Breast cancer-specific survival is defined as the time from inclusion to death from breast cancer.
Overall survival (OS) | From date of beginning of hormonotherapy to death from any cause, up to 10 years.
  The overall survival is the length of time from inclusion to death from any cause.
Quality of life (QoL) questionnaire - Core 30 (QLQ-C30) | At baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life (QoL) questionnaire - EORTC QLQ-BR23/QLQ-BR45 | At baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR23 contains 23 items incorporating five multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning. In addition, single items assess sexual enjoyment, hair loss and future perspective. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. For all items but sexual functioning and sexual enjoyment, higher scores indicate more severe symptoms. The QLQ-BR-23 was updated and 22 new questions were added to provide a more accurate and comprehensive assessment of the impact of new and scalable treatments on patients'QoL
Quality of life (QoL) questionnaire - Cancer related fatigue (QLQ-FA12) | At baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  This EORTC cancer related fatigue questionnaire is intended to supplement the QLQ-C30.
  The QLQ-FA12 contains 12 items organized in three subscales: physical fatigue (5 items), emotional fatigue (3 items), and cognitive fatigue (2 items). The remaining two items serve as global indicators for interference of fatigue with daily activities and social sequelae of fatigue.
  All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale with higher scores indicating greater degree of fatigue.
Hospital anxiety and depression scale (HADS) | At baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  The HADS is a 14 items questionnaire: 7 items related to anxiety and 7 items related to depression scored on a scale. Scores for items in each subscale of the HADS are summed to produce an anxiety score (HADS-A) or a depression score (HADS-D), or can be added to produce a total score corresponding to emotional distress (HADS-T). Each item is rated on a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), for a total score ranging from 0-21 for each subscale. The entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress.
Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) | At baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  The FACT-Cog is a self-assessment questionnaire to estimate memory, attention, concentration, language, and thinking abilities of patients before, during, and after chemotherapy. This questionnaire, composed of 37 items consists of four subscales: cognitive impairments perceived by the patient (20 items), comments from others (4 items), cognitive abilities perceived by the patient (9 items), and impact on quality of life (4 items). The Perceived Cognitive Impairments and the Comments from Others subscales are rated on 5-point Likerttype scale (from 0 = "Never" to 4 = "Several times a day"). An intensity 5-point Likert-type scale (from 0 "Not at all" to 4 "Very much") is used to rate perceived cognitive abilities and the impact on quality of life. For all subscales, a higher score represents better cognitive functioning or quality of life.
Impact of Cancer (including fear of recidivism) | At baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  The Impact of Cancer Version 2 (IOCv2) is a 47-item questionnaire. The first 37 items are intended to measure 4 positive (Altruism/Empathy, Health Awareness, Meaning of Cancer, and Positive SelfEvaluation) and 4 negative (Appearance Concerns, Body Change Concerns, Life Interferences, and Worry) subscales, which total to two summary scores (Positive and Negative Impact). The 10 additional items constitute conditional dimensions applicable to subsets of survivors assessing employment concerns, relationship concerns for individuals with a partner, and relationship concerns for those without a partner. All items are scored on a five-point scale (1 = "strongly disagree", 2 = disagree, 3 = neutral, 4 = agree, and 5 = "strongly agree"). Higher scores on the positive impact indicate greater positive impacts, while higher scores on the negative impact indicate greater negative impacts.
Geriatric Core Dataset (G-CODE) | At baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  The G-CODE was developed by the DIalog for personALization of management in geriatric OncoloGy (DIALOG) intergroup to assess the general health status of the older patient.
  The G-Code contains 10 tools incorporating seven scales to assess social environment, functional status, mobility, nutritional status, cognitive status, depressive mood, and comorbidities. The total scale range 0-62. High score indicate better condition.
Evaluate the safety of the treatment in the study population | Throughout study completion, up to 10 years.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5.0) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Elise DELUCHE, MD, Study Chair — CHU Limoges; Fabrice André, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Institute Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No